CLINICAL TRIAL: NCT04649762
Title: Evaluation of the Activating Consciousness Technique (Hypnosis) in Anxiety in a General Practice
Brief Title: the Activating Consciousness Technique (Hypnosis) in General Practice
Acronym: MG HYPNOSIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0202
Record Dates: First submitted 2020-09-29; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Anxiety
Keywords: hypnosis; anxiety; general practice
MeSH Terms: conditions — Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Group 1 includes patients with anxiety consulting a doctor not practicing hypnosis
- TAC: Group 2 includes patients with anxiety consulting a doctor practicing hypnosis
  Interventions: Behavioral: activating consciousness technique (hypnosis)

INTERVENTIONS:
Behavioral: activating consciousness technique (hypnosis) — activating consciousness technique (hypnosis)
  Groups: TAC

SUMMARY:
Anxiety is an emotion considered unpleasant but resulting from a normal phenomenon. It corresponds to an adaptive response to events, to stress and helps to ensure our survival.

On the other hand, it becomes embarrassing when it becomes uncontrollable. It can even lead to interfere with activities of daily living. Thus, we can speak of anxiety disorder.

Anxiety disorders are among the most prevalent psychiatric disorders. They are often associated with other comorbidities such as depression, which makes them more difficult to treat and diagnose.

Different treatments are offered to best treat the patient with anxiety : drug treatment (antidepressants, anxiolytics) ; non-drug (psychotherapy, meditation, cognitive behavioral therapies).

The emergence of hypnosis in medical practice in recent years seems to be a technique that can bring benefits to the patient.

A review of clinical studies does not seem to find a benefit to hypnosis in anxiety disorders. In contrast, a study in children with school phobia showed the effectiveness of hypnosis. The limits addressed by this review seem to relate to the number of people included in the studies. Contrariwise, it has been pointed out that hypnosis can have a beneficial effect in the long term.

Thus, it seems interesting to deepen this technique in the practice of a general practitioner exercising the activating consciousness technique in anxiety.

The study will be composed of patients presenting with anxiety and consulting their general practitioner, with: Group 1, patients consulting a doctor not practicing hypnosis Versus Group 2, patients consulting a doctor practicing hypnosis.

During the first consultation and the following 2 consultations scheduled by the general practitioner (spaced 15 days apart), the following data are noted, in addition to the monitoring usually performed by the doctor:

1. COVI scale
2. Comfort scale 0 to 10
3. Management: drugs, TAC, others
4. Quality of life survey SF36 Patients will be called back at 6 months to reassess quality of life (self-administered survey SF 36) The primary endpoint is to evaluated the change of anxiety from inclusion (J0) to 6 months using COVI scale in the two different groups.

For secondary endpoints, the consumption of drug medicine will be quantified and the quality of life will be measured using Quality of life survey SF36.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18
* Anxiety patient
* Patient who can return for consultation regularly and can be reached by phone
* Patient Not Opposing Participation In Study

Exclusion Criteria:

- Follow-up deemed impossible by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with anxiety according to DSM V-C criteria: 3 of 6 symptoms
  * Agitation or sensation of being overflown or exhausted
  * Fatigability
  * Difficulty concentrating or memory lapses
  * Irritability
  * Muscle tension
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change of the score of anxiety from inclusion (J0) to 6 months evaluated byvia COVI scale | 6 months
  COVI scale (questionnaire completed by patients) is a scale that permits to evaluate the clinical anxiety. The range is 0-100. The higher the score, the more the anxiety. The clinical cut-off score is 30.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Dr Stéphane FOLACHER, Bourg-en-Bresse
  - Dr Céline HUMBERT, Lyon
  - Dr Matthieu DEMOURGUES, Lyon
  - Dr Christian SAINT-CYR, Saint-Étienne-du-Bois
  - Dr Aurélien BARADEL, Saint-Martin-du-Frêne
  - Dr Maud BINARD, Villereversure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelissolo A. [Hypnosis for anxiety and phobic disorders: A review of clinical studies]. Presse Med. 2016 Mar;45(3):284-90. doi: 10.1016/j.lpm.2015.12.002. Epub 2016 Mar 2. French. PMID 26944812